CLINICAL TRIAL: NCT05378126
Title: Prospective Pilot Study Evaluating the Prognostic Impact of a Neuro-vascular Examination Associated with Cerebral MRI in the Acute Phase of Infectious Endocarditis
Brief Title: Evaluation of the Prognostic Impact of a Neuro-vascular Examination Associated with Cerebral MRI in the Acute Phase of Infectious Endocarditis
Acronym: POMPEI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL18_0798
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Endocarditis; Stroke
Keywords: Neurological assessment; Medical care
MeSH Terms: conditions — Endocarditis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neurological cohort (Other): All patients included in the study wil have a neurological examination
  Interventions: Other: Neurological assessment

INTERVENTIONS:
Other: Neurological assessment — No specific procedure is planned for the study other than the neurological examination by a neurologist of all patients. The patient will be taken care according to current recommendations.
  In addition, a study-specific, non-injected brain CT scan will be performed systematically in patients undergoing cardiac surgery to evaluate postoperative hemorrhagic transformation.

SUMMARY:
Infectious endocarditis (IE) is a serious condition with an annual incidence of 3 to 10 per 100,000 people. Brain infarctions complicate approximately 20-40% of endocarditis.

Brain MRI can detect the presence of recent ischemic lesions and asymptomatic microbleeds. Preoperative brain imaging is part of the recommended assessment in the management of IEs, but the type of imaging and sequences are not codified and the impact of cerebral and vascular imaging findings on the therapeutic decision remains uncertain.

The level of evidence of the recommendations remains low, especially for complicated IEs of stroke. There is very little neurological clinical data on patients with IEs. Similarly, neurologists do not systematically participate in multidisciplinary meetings during the management of an IE. It therefore seems interesting to carry out a neurological cohort of this population and to evaluate what would be the contribution of vascular neurologists in the management of infectious endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Certain infectious endocarditis according to Dukes Criteria
* Signed informed consent

Exclusion Criteria:

* Hospital admission due to neurovascular emergency
* MRI contraindications
* Pregnant or women of childbearing age who were not using contraception (oral diagnosis),
* Patient without health coverage,
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Medical care modification | at 3 months
  Description of the medical care modification after neurological assessment, evaluated by the number of patients with modified medical care by the request for a new examination compared to the initially scheduled care.
Medical care modification | at 3 months
  Description of the medical care modification after neurological assessment, evaluated by the number of patients with modified medical care by the change of therapy compared to the initially scheduled care.

SECONDARY OUTCOMES:
The description of the preoperative neurological impairment | During initial hospitalization
  Description of preoperative neurological impairment assessed by NIHSS score
The description of the preoperative neurological impairment | During initial hospitalization
  Description of preoperative neurological impairment assessed by the presence of brain lesions on initial MRI
The description of the perioperative hemorrhagic risk | 24 to 96 hours post-surgery
  Description of the perioperative hemorrhagic risk evaluated by the rate of haemorrhagic transformation on the post-surgery control scanner
Prognosis assessment | at 3 months
  Evaluation of prognosis by the rate of deaths and stroke
Evaluation of functional prognosis | at 3 months
  Evaluation of the functional prognosis measured by the mRS score
Evaluation of depressive anxiety disorders | at 3 months
  Evaluation of depressive anxiety disorders measured by the Hamilton Anxiety Depression scale
Evaluation of the cognitive prognosis | at 3 months
  Evaluation of the cognitive prognosis evaluated by the MOCA score

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Unit, Pierre Wertheimer hospital, GHE Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No